CLINICAL TRIAL: NCT04102228
Title: A Randomized Sham-Controlled Trial of Repetitive Transcranial Magnetic Stimulation (rTMS) and Multi-Modal Aphasia Treatment (M-MAT) for Post-Stroke Non-Fluent Aphasia
Brief Title: Repetitive Transcranial Magnetic Stimulation and Multi-modality Aphasia Therapy for Post-stroke Non-fluent Aphasia
Acronym: REMAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Sean Dukelow, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB19-0829
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Stroke; Aphasia, Non-fluent
Keywords: Non-invasive brain stimulation; Transcranial Magnetic Stimulation; Multi-modality aphasia therapy; Neuroimaging
MeSH Terms: conditions — Stroke; Aphasia, Broca

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups for the duration of the study (Multi-modality aphasia therapy plus inhibitory rTMS or multi-modality aphasia therapy plus sham rTMS).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-modality aphasia therapy plus 1Hz rTMS (Experimental): Participants receive 10 days of 3.5hrs of multi-modality aphasia therapy (M-MAT) preceded by 20 minutes of 1Hz rTMS delivered at 100% of resting motor threshold over the right pars triangularis.
  Interventions: Device: 1Hz inhibitory rTMS; Behavioral: Multi-Modality Aphasia Therapy (M-MAT)
- Multi-modality aphasia therapy plus sham rTMS (Sham Comparator): Participants receive 10 days of 3.5hrs of multi-modality aphasia therapy (M-MAT) preceded by 20 minutes of sham rTMS is achieved using a sham TMS coil which attenuates the magnetic output of the stimulator by 80%.
  Interventions: Device: 1Hz sham rTMS; Behavioral: Multi-Modality Aphasia Therapy (M-MAT)

INTERVENTIONS:
Device: 1Hz inhibitory rTMS — 20 minutes of 1Hz (1200 pulses) repetitive transcranial magnetic stimulation (rTMS) applied by Magstim Rapid 2 stimulator equipped with an airfilm figure-8 coil
  Arms: Multi-modality aphasia therapy plus 1Hz rTMS
Device: 1Hz sham rTMS — 20 minutes of 1Hz (1200 pulses) repetitive transcranial magnetic stimulation (rTMS) applied by Magstim Rapid 2 stimulator equipped with an airfilm figure-8 sham coil.
  Arms: Multi-modality aphasia therapy plus sham rTMS
Behavioral: Multi-Modality Aphasia Therapy (M-MAT) — Participants receive 3.5 hours of intensive speech therapy in small groups delivered by a blinded speech language pathologist and therapy assistant. The objective of M-MAT is to improve word production through shaping of responses (ie. Gradually increasing complexity of spoken targets towards eventual mastery) and social-mediated repetitive practice. Therapists use game-based interactive tasks and rich multi-modal cueing (gestures, written words, drawing, reading words) to improve spoken production and oral communication.

SUMMARY:
Many stroke survivors experience aphasia, a loss or impairment of language affecting the production or understanding of speech. One common type of aphasia is known as non-fluent aphasia. Patients with non-fluent aphasia have difficulty formulating grammatical sentences, often producing short word fragments despite having a good understanding of what others are trying to communicate to them. Speech language pathologists (SLPs) play a central role rehabilitating persons with aphasia and administer therapy in an attempt to improve communication skills. Despite standard therapy, approximately 50% of individuals who experience aphasia acutely continue to have language deficits more than 6 months post-stroke.

In most people, Broca's area is dominant in the left side of the brain. Following a left-sided stroke, the right-sided homologue of Broca's area (the pars triangularis), may adopt language function. Unfortunately, reorganizing language to the right side of the brain seems to be less effective than restoring function to the left hemisphere. Repetitive transcranial magnetic stimulation (rTMS), a form of non-invasive brain stimulation, can be used to suppress activity of specific regions in the right side of the brain to promote recovery of function in the perilesional area. Despite preliminary success in existing studies using rTMS in post-stroke aphasia, there is much work to be done to better understand the mechanisms underlying recovery. Responses to rTMS have been positive, yet heterogenous, which may be related to timing of treatments following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Isolated left middle cerebral artery (MCA) stroke within past 6 months (sub-acute) or more than 6 months ago (chronic)
* Stroke type: Ischemic or hemorrhagic
* Non-fluent aphasia as determined by the Western Aphasia Battery (Fluency < 5)
* English is first or primary language
* Ability to follow 3-step commands

Exclusion Criteria:

* Prior stroke to the right frontal lobe
* Current diagnosis of moderate to severe depression
* Diagnosis of any other psychiatric condition
* History of other neurologic disorders (e.g., epilepsy, brain tumor)
* Contraindication to MRI or TMS (metal in the head or any implanted electrical device)
* Has received intensive speech therapy within the past 6 months (>8 hours per week)
* Enrolled in another interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the Western Aphasia Battery (Revised) Aphasia Quotient within one week of intervention completion | Baseline, within 1 week of completing the 10 day intervention
  Western Aphasia Battery Aphasia quotient (WAB-AQ) composite score, composed of fluency, spontaneous speech, naming, and comprehension sub-tests. Scores range from 0 to 100, with higher scores indicating better overall speech and language abilities. Positive change from baseline indicates better outcome.
Change from baseline on the Western Aphasia Battery (Revised) Aphasia Quotient at 3 months | Baseline and 3-month follow-up
  Western Aphasia Battery Aphasia quotient (WAB-AQ) composite score, composed of fluency, spontaneous speech, naming, and comprehension sub-tests. Scores range from 0 to 100, with higher scores indicating better overall speech and language abilities. Positive change from baseline indicates better outcome.

SECONDARY OUTCOMES:
Trained and Untrained Picture Naming | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Number of correctly named pictures from a set of trained nouns, trained verbs, untrained nouns, and untrained verbs.
Scenario Test (UK) | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Test of functional communication based on everyday conversational scenarios
Connected speech sample | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Records the number of correct information units provided by participants while re-telling a familiar story (e.g., the three little pigs)
Cognitive Linguistic Quick Test - aphasia administration | Baseline
  Brief assessment of non-verbal cognition
Overt Naming Functional Magnetic Resonance Imaging | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Functional neuroimaging collected during picture naming task to assess activity associated with naming
Resting-state Functional Magnetic Resonance Imaging | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Functional neuroimaging collected during rest to be used for functional connectivity
Magnetic Resonance Spectroscopy | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  1H proton spectroscopy used to measure metabolite concentrations within the right inferior frontal gyrus
Diffusion weighted Magnetic Resonance Imaging | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Neuroimaging measuring the diffusion of water to be used for white matter reconstruction
Communication Effectiveness Index | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Caregiver completed questionnaire to assess functional communication
Stroke Aphasic Depression Questionnaire (SADQ) | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  A 10-item questionnaire completed by a caregiver to quickly assess depressive symptoms in stroke patients with aphasia.
Stroke and Aphasia Quality of Life Scale (SAQOL) | Baseline, within 1 week of completing the 10 day intervention and 3-month follow-up
  Assesses mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ also records the patient's self-rated health on a vertical visual analogue scale. This can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Western Aphasia Battery - Bedside (WAB) | Screening appointment
  Assesses the linguistic skills and main nonlinguistic skills of adults with aphasia. This provides information for the diagnosis of the type of aphasia.
Apraxia Battery for Adults (ABA) | Screening appointment
  Assesses characteristics of verbal apraxia

CONTACTS AND LOCATIONS:
Overall Officials: Sean P Dukelow, MD PhD FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers

REFERENCES:
- [Derived] Low TA, Lindland K, Kirton A, Carlson HL, Harris AD, Goodyear BG, Monchi O, Hill MD, Rose ML, Dukelow SP. Transcranial Magnetic Stimulation Combined With Multimodality Aphasia Therapy for Chronic Poststroke Aphasia: A Randomized Clinical Trial. Neurology. 2025 Mar 25;104(6):e213424. doi: 10.1212/WNL.0000000000213424. Epub 2025 Feb 25. PMID 39999397

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT04102228/SAP_000.pdf